CLINICAL TRIAL: NCT05426863
Title: Integrated Multicomponent Intervention for Violence Prevention and Management of Mental Health Problems Among Women Experiencing IPV in Madhesh Province of Nepal: A Cluster Randomized Trial.
Brief Title: Domestic Violence Intervention to Reduce Psychological Distress and Violence Among Women Experiencing IPV in Nepal
Acronym: DeVI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Global and Sexual Health (GloSH) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 555
Record Dates: First submitted 2022-06-08; First posted 2022-06-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Intimate Partner Violence; Domestic Violence; Intervention; Mental Health; Secondary Prevention; Problem Management Plus; Cluster Randomized Trial
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Psychosocial Counselling (Experimental): A multi-component intervention counseling package to prevent the reoccurrence of IPV and address psychological distress among women experiencing violence. The DeVI intervention is structured into five weekly sessions.
  Interventions: Behavioral: DeVI
- Standard Usual Care (No Intervention): Provide standard usual care and information booklet similar to that of the intervention group that contains updated contact information for the referral services.

INTERVENTIONS:
Behavioral: DeVI — A multi-component intervention is devised from the components of PM+ developed by WHO incorporating the components of violence prevention. The intervention is anticipated to provide behavioral skills to the participants in the intervention arm which will enhance their coping skills with past experiences of violence, stress management skills, problem-solving skills and safety planning skills. Further, they will be shared the best practices and lessons learned which will aid in danger assessments and prevention of future violence. The intervention will be given to intervention arm in 5 different sessions, one in each week. The 1st session of the intervention is about understanding the multi-component intervention. The 2nd session is identifying and managing problem, 3rd session is about stress management, followed by development of safety plan in 4th session and last session is about promotion of social support.
  Arms: Psychosocial Counselling

SUMMARY:
The aim of this study is to implement and evaluate the feasibility, acceptability, and effectiveness of a validated integrated multi-component intervention targeting secondary prevention of violence and addressing the mental health needs of women experiencing intimate partner violence.

DETAILED DESCRIPTION:
This study's aim is to assess the feasibility and effectiveness of an integrated multicomponent intervention among women experiencing violence in Madhesh Province of Nepal.

1. To assess the feasibility of DeVI in health care centers in Nepal by exploring the views of key stakeholders, health care providers, and local women in the community.
2. To train non-specialist mental health care providers on the delivery of DeVI among women exposed to IPV.
3. To explore participants' and health care providers' experiences with DeVI Intervention and the opportunities and challenges encountered during implementation.
4. To measure the effectiveness of the DeVI intervention in addressing psychological distress, reducing the occurrence of IPV, and developing safety strategies among women experiencing IPV.
5. To measure the impact of the DeVI training on knowledge, attitudes, skills, and stigma towards IPV and its consequences, particularly on psychological trauma among health care providers.

ELIGIBILITY:
Inclusion Criteria:

* Women between the age of 18-49 years
* Having experienced abuse (physical, sexual, or psychological) in a heterosexual relationship from her husband or her family members in the last 12 months
* Non-pregnant or pregnant in the first trimester
* Score of 3 and above in the psychological distress scale (measured by General Health Questionnaire (GHQ-12))
* Living with her husband or in-laws for at least six months.

Exclusion Criteria:

* Have a severe cognitive impairment
* Seeking treatment for life-threatening emergency care
* Have suicidal thoughts

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 912 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2024-02-22 (Actual)

PRIMARY OUTCOMES:
General Health Questionnaire (GHQ-12) | Baseline Assessment (T1); Changes from Baseline assessment, at 1 week post-intervention assessment (6 weeks after Baseline) (T2), Changes from Baseline assessment, at 12 week post-intervention assessment (17 weeks after Baseline) (T3)
  12 item measures for psychological disorders in non-clinical settings, minimum value=0 maximum value=12; higher scores mean greater distress
Intimate partner violence or domestic violence | Baseline(T1),Changes from Baseline, at 1 week post-intervention(6 weeks after Baseline)(T2),change from baseline, at 12 week post-intervention(17 weeks after Baseline) (T3),Changes from Baseline,at 47 week post intervention(52 weeks after baseline) (T4)
  We will document the change in the experience of IPV or domestic violence using modified WHO multi country questionnaire. Defined as violence in the different time frame with participants' husband/male partner/ in-law's. a) Controlling behaviors: "presence of at least one behavior (restrict contact with participants family of birth, ignore participants and treat indifferently etc.)". b) Psychological violence: "insulted participants to made participant's feel bad about herself, belittled or humiliated you in front of other people, yelling and smashing things to scare participants, threat to hurt participants or her close one". c) Physical violence: "slapped, pushed or pulled; hit with fist or something else; kicked, dragged or beating; choked or burnt on purpose; threatened with gun, knife or other weapon". d) Sexual violence: "physically forced participants to have sexual intercourse; forced to do something sexual that is degrading or humiliating etc."

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | Baseline(T1),6 weeks after Baseline(T2), 17 weeks after Baseline(T3)
  9-item measure of depression symptoms; minimum value = 0, maximum value = 27; higher scores mean more severe depression symptoms support, impaired functioning, symptoms of post-traumatic stress, personally identified problems, and health service utilization.
Post-traumatic stress Disorder (PTSD)-(PCL-C) | Baseline(T1), 6 weeks after Baseline(T2), 17 weeks after Baseline(T3)
  17-item measure of Post-traumatic stress disorder; minimum value=17 maximum value=85. The 17-29=little to No PTSD symptoms, 28-29=some PTSD symptoms, 30-44=moderate severity of PTSD symptoms and 45-85 =high severity of PTSD symptoms.
The Hospital Anxiety and Depression Scale (HADS) | Baseline(T1), 6 weeks after Baseline(T2), 17 weeks after Baseline(T3)
  Measure of anxiety disorders and depression; minimum value=0 maximum value=21. 7 or less indicate non anxiety and non-depression cases, 8 to 10 indicates borderline cases, 11 and above indicates definite cases.
Perceived Social Support | Baseline(T1), 6 weeks after Baseline(T2), 17 weeks after Baseline(T3)
  5-items measures of support received from the community; minimum value=5 (less perceived support) maximum value=25(higher perceived support)
WHO Disability Assessment Schedule (WHODAS 2.0) | Baseline(T1), 6 weeks after Baseline(T2), 17 weeks after Baseline(T3)
  12-items measure of difficulties of individual in performing the certain activities; minimum value=0 maximum value=48
PSYCHLOPS | Baseline(T1), during intervention (in intervention arm only), 6 weeks after Baseline(T2), 17 weeks after Baseline (T3)
  Measures of the problem and its effect in wellbeing and daily functioning over the last week; minimum value=0 maximum value=20 higher score denotes higher severity of psychological stress and functioning.
Safety Behaviour Checklist and Use of Community Resource | Baseline(T1), 6 weeks after Baseline(T2), 17 weeks after Baseline(T3), 52 weeks after Baseline (T4)
  Measure the safety measures adopted by the participants in advance of potentially dangerous situations; the utilization of the local services available in the community for the prevention or the reduction of the violence occurrence
Modified Physical Readiness to Manage IPV Survey (PREMIS) | Immediately after Integrated multi component Intervention Training (10 days post -baseline), during Integrated multicomponent supervision (approximately 90-days post-baseline)
  7-items measures of actual IPV knowledge, 23-items measures of attitude towards IPV, and 10-items measures of practice issues. All these items will be presented in descriptive format i.e. frequency and percentage of each option of each question selected by participants.
Mental Health knowledge Schedule (MAKS) | Immediately after Integrated multi component Intervention Training (10 days post -baseline, during Integrated multicomponent supervision (approximately 90-days post-baseline)
  MAKS consists of six stigma-related mental health knowledge areas; employment, recognition, treatment, supports, help-seeking and recovery and knowledge and mental health conditions. MAKS comprises 12 items; among which 4 are negative statements. Each item has 5 points Likert scale score ranging from 1-5. For the positive statement, 'Strongly Agree' scores the highest 5 points, whereas 'Strongly Disagree' scores 1. The points in the ordinal scale are reversed for the negative statements. The totals score is calculated summing up the score of each of the 12 items. Higher score indicates higher participant's knowledge on mental health. We will document the change in the mean scores of mental health literacy between the two arms measured using MAKS.
Social Distance Scale | Immediately after Integrated multi component Intervention Training (10 days post -baseline)
  Social Distance Scale is aimed for the healthcare providers to measure their attitude towards the people with mental health. It is 7-item scale consisting 4 points scale each item ranging between 0-3, where 0 = definitely willing, 1= willing, 2= unwilling and 3 = definitely unwilling. Possible scores thus range from 0 to 21, with higher scores representing a greater desire to distance oneself from persons who have mental illness.
Perceived Dangerousness of the Mental Health Patients | Immediately after Integrated multi component Intervention Training (10 days post -baseline)
  Perceived Dangerousness scale measures will be used to assess the perceived perceptions of health workers towards mental health patients. The scale consists of 8 items and responses on each item were measured using a six-point scale 0-5; ranging from strongly agree-strongly disagree. Majority of the statements are negative with reversed options order. The total score ranges from 0-40. The score will be obtained in each item by summing up to obtain a total score, which is divided by eight to create a scale varying from 0-5. The high score reflects the belief / perception that the people with mental illness are dangerous.

OTHER OUTCOMES:
Exit Client Interview | at 1 week post-intervention assessment (T2)
  Exit client interview will be used to measure satisfaction and acceptability of the intervention from the participant's point of view in the intervention arm. A total of 15 mixed qualitative and quantitative questions will be used. Quantitative questions ranges from 0-17, higher scores means both satisfied and accepted intervention while lower score means not satisfied and not accepted the intervention. In addition qualitative question will be asked to understand and know more about the satisfaction and acceptability of intervention among the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Keshab Deuba, PhD, Principal Investigator — Karolinska Instituet
Locations (1):
- DeVI Intervention Site, Janakpur Dham, Madhesh, Nepal

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual data will be available through K2A Data Archive after publication of primary results.
Supporting Information: Study Protocol, ICF
Time Frame: Materials will be shared after publication of primary results.
Access Criteria: Contact PI.

REFERENCES:
- [Derived] Shrestha R, Sapkota D, Mehra D, Ekstrom AM, Deuba K. Feasibility and Effectiveness of an Intervention to Reduce Intimate Partner Violence and Psychological Distress Among Women in Nepal: Protocol for the Domestic Violence Intervention (DeVI) Cluster-Randomized Trial. JMIR Res Protoc. 2023 Aug 15;12:e45917. doi: 10.2196/45917. PMID 37581909